CLINICAL TRIAL: NCT05358392
Title: "Effect of Emotional Freedom Technique Application on Infertility Stress in Women"
Brief Title: "Effect of Emotional Freedom Technique "
Acronym: (EFT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonca Karatas Baran (Other)
Responsible Party: Sponsor-Investigator, Gonca Karatas Baran, Dr Nurse, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Organization: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Etlik SagBakHizm
Record Dates: First submitted 2022-04-21; First posted 2022-05-03 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Emotions; Infertility; Stress
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Since there is no reference study on this subject, the effect width will be calculated for the main research question by making a preliminary application (9 cases, 9 controls) and the sample will be calculated with 90 power and 0.05 margin of error in the effect width obtained. Block randomization (3 blocks as male infertility, female infertility and unexplained infertility) for the pre-application intervention and control groups was performed through the Randomization Sofcare Allocation program. In the main application, this program will be made according to the number of samples and the intervention and control groups will be assigned. Pre-application data will be included in the research analysis.
  The Patient Follow-up Form consists of 3 parts. In the first part, there are data on socio-demographic and obstetric characteristics. The second part includes the infertility stress scale (pre-test) and the third part includes the infertility stress scale (post-test).
Who Masked: Participant
Masking Description: : Women who applied to Etlik Zübeyde Hanım Gynecology Training and Research Hospital IVF/ICSI unit for IVF/ICSI treatment. who meet the criteria for inclusion in the study will be informed about the study, and the women who accept the study will be assigned to the groups determined by randomization.After participating in the study, the participants will know which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- emotional freedom technique (Experimental): 5 sessions of EFT* will be applied to this group on the first day of the treatment, 1st Control, 2nd Control, before the OPU procedure and before the embryo transfer. Subjective discomfort level will be measured with SUD** before and after each application.
  Interventions: Other: emotional freedom technique (EFT)
- control (No Intervention): No application will be made to this group. Infertility stress scale will be filled in the case and control group at the beginning of the treatment and after the embryo transfer.

INTERVENTIONS:
Other: emotional freedom technique (EFT) — EFT is an energy psychotherapy derivative application, consisting of cognitive and somatic components, used to heal personal negative emotions and related emotional and physical disorders. Stress hormones are secreted in response to the stress response in the person, and then the amygdala and other cerebral parts that respond to stress are activated. There are basic steps to be followed in EFT application; By giving a message to the emotional body (subconscious) with suggestion sentences, clicks are made on the twelve energy meridian endpoints (acupressure points).
  Arms: emotional freedom technique

SUMMARY:
This study will be conducted to investigate the effect of Emotional Freedom Technique (EFT) Application on infertility stress in women undergoing infertility treatment.

DETAILED DESCRIPTION:
Emotional Freedom Technique (EFT) is an easy-to-apply therapy, one of the types of energy psychotherapy. EFT gives effective and successful results in clinical problems.

Personal energy level and balance are very important, as Gary Craig, the inventor of the technique, stated, "The cause of all negative emotions is due to the disorder in the body's energy system." Because any disruption or blockage in the energy flow brings with it physical and psychological disorders. For this reason, first of all, the negative emotion that causes the negative situation should be eliminated. When the energy flow in the meridians is balanced, the emotional intensity or negative/negative emotion also disappears. Thus, the person starts to feel good.

In energy psychology applications, while the individual is in a relaxed and relaxed state, the electrical energy flow in the meridian system is also comfortable and regular. Emotional reactions such as anger, sadness, stress, disappointment create sudden obstacles in this flow. By focusing on the emotional reactions that hinder the individual, the stimulations on the meridian system (often by touch) regulate the energy flow and provide the individual to relax. The fact that the flow in the meridian system is not interrupted provides relief in the mind, body and emotion areas of the individual.

EFT works on the cognitive and energetic levels. While it is ensured that the individual is conscious and aware of a disturbing symptom or disorder, selected acupuncture points are touched at the same time, creating a cognitive transition and energetic release. EFT is applied safely for stress management.

It can be safely applied to individuals of all ages, including the elderly, pregnant and children. EFT was applied in 51 studies, 18 of which were randomized controlled and positive results were obtained with clinical measurements.

With EFT, the energy flow can be regulated safely and consciously, contributing to the individual's "better" feeling. Positive results in past applications reveal the reliability of the method. Since the application procedure is easy, the application areas are versatile and it does not show side effects, it is recommended that EFT be widespread in different clinical areas and evidence-based studies should be increased.

ELIGIBILITY:
Inclusion Criteria:(For the intervention and control group):

* Women who have applied to the IVF clinic for primary infertility treatment,
* in the initial stage of IVF/ICSI treatment,
* literate in Turkish,
* have no chronic disease,
* have no diagnosed psychiatric disease,
* between the ages of 18-40,
* agree to participate in the study.

Exclusion Criteria:

* Women with a diagnosis of secondary infertility who do not meet the conditions for inclusion in the study (for the intervention and control group),
* Women want to leave the study (for the intervention group) before the implementation phases are completed.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
INFERTILITY STRESS SCALE score | change from baseline ınfertility stress scale score ( approximately 15 days later ınfertility treatment)
  This scale, which will be applied to evaluate the stress experienced by infertile women.The scale has three sub-dimensions related to "personal", "marriage" and "social" fields and consists of 14 items in total.

SECONDARY OUTCOMES:
Subjective Level of Discomfort | 1,2,3,4,5. times EFT ıntervention (First 15 days of ınfertility treatment)
  It is the subjective rating of discomfort felt by the patient. Before starting the application in energy therapies, it is requested to evaluate the severity of the discomfort caused by the problem on a graded measurement called Subjective Units of Disturbance-SUD, which was used by Wolpe before. During this subjective evaluation, the client considers the discomfort he feels as 10 unbearable discomfort, 0 no discomfort, and scores it on a scale of 0-10. By means of this scoring, the severity of the discomfort felt by the individual at that moment is determined.
pregnancy status (positive or negativity according to BHCG value) | 30 days later of ınfertility treatment
  BHCG value evaluation in the blood (routinely applied in those who have ınfertility treatment)

CONTACTS AND LOCATIONS:
Overall Officials: GONCA K KARATAS BARAN, PHD, Principal Investigator — Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Locations (1):
- Gonca Karataş Baran, Ankara, Eyalet/Yerleşke, Turkey (Türkiye)